CLINICAL TRIAL: NCT06200844
Title: The Efficacy of Three Doses of Live Attenuated, Oral Rotavirus Vaccine 116E (ROTAVAC 5D) in Chilean Infants.
Brief Title: The Efficacy of Oral Rotavirus Vaccine 116E (ROTAVAC 5D) in Chilean Infants
Acronym: Rota5DCHILE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BBIL/Rotavac 5D-CHILE /2022
Record Dates: First submitted 2023-12-11; First posted 2024-01-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Rotavirus Infection of Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rotavac 5D (Experimental): Rotavirus Vaccine (ROTAVAC 5D), is a monovalent vaccine containing suspension of live attenuated rotavirus 116E prepared in Vero cells, containing NLT 10 power 5.0 FFU and administered as a three-dose regimen, 4 weeks apart.
  Interventions: Biological: ROTAVAC 5D
- Placebo (Placebo Comparator): Placebo administered as a three-dose regimen, 4 weeks apart.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ROTAVAC 5D — Rotavirus Vaccine (ROTAVAC 5D), is a monovalent vaccine containing suspension of live attenuated rotavirus 116E prepared in Vero cells, containing NLT 105.0 FFU and administered as a three-dose regimen, 4 weeks apart.
  Arms: Rotavac 5D
Other: Placebo — Placebo is administered as three doses 4 weeks apart
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, phase 3 study to evaluate the Efficacy,Safety, and Immunogenicity of ROTAVAC 5D, a live attenuated rotavirus vaccine in healthy infants aged 6-8 weeks.

A total of 5800 healthy Chilean infants will be recruited in this study and randomized to receive either vaccine or placebo in 1:1 ratio. Among these participants 300 will be categorized to immunogenicity cohort, 150 from each group, and blood samples will be collected to assess the immune response.

DETAILED DESCRIPTION:
The Efficacy of Three Doses of Live Attenuated, Oral Rotavirus Vaccine 116E (ROTAVAC 5D) in Chilean Infants.

This is a randomized, double-blind, phase 3 study to evaluate the Efficacy, Safety, and Immunogenicity of ROTAVAC 5D, a live attenuated rotavirus vaccine in healthy infants aged 6-8 weeks.

A total of 5800 healthy Chilean infants will be recruited in this study and randomized to receive either vaccine or placebo in 1:1 ratio. Among these participants 300 will be categorized to immunogenicity cohort, 150 from each group, and blood samples will be collected to assess the immune response. Inclusion At least one parent(s) or legally acceptable representative's consent for participation and are able to understand study procedures Subjects aged 6 to 8 weeks at recruitment No plans to move in the next 12 months Exclusion Administration of rotavirus vaccine in the past Presence of any illness requiring hospital referral (temporary exclusion) Known case of immunodeficiency disease, known HIV positive Known case of chronic gastroenteritis disease, chronic pulmonary disease, chronic renal disease, congenital heart disease Any other conditions which in the judgment of the investigator warrant exclusion (e.g. no exclusion criteria but seems 'ill', investigators suspects neglect) Diarrhea on the day of enrollment (temporary exclusion) A known sensitivity or allergy to any components of the study vaccines. Major congenital or genetic defect. Has received any immunoglobulin therapy and/or blood products since birth. History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study, at the discretion of the principal investigator. Blood samples: In the "Immunogenicity Subset", 3 ml blood specimens will be collected at baseline and 28 (+) 5 days after the third dose of the Test Article/placebo to assess the anti rotavirus IgA antibody titer. Stool Specimens: The study team will attempt to collect a stool specimen for every GE episode, preferably within the first 2 days after episode onset. The stool specimen may be collected up to 7 days after the last day of diarrhea. The stool specimens will be sent to the laboratory. If the episode is a suspected intussusception or vaccine associated gastroenteritis that has occurred within four weeks after each dose of the Test Article/placebo, the specimen will be sent to the laboratory immediately for rotavirus testing and typing. For all ELISA RV positive samples, an aliquot of the stool specimen will be assessed for 20 enteropathogens by multiplex-PCR panel and to identify the genotype of the virus.

ELIGIBILITY:
Inclusion Criteria:

1. At least one parent(s) or legally acceptable representative's consent for participation and are able to understand study procedures
2. Subjects aged 6 to 8 weeks at recruitment
3. No plans to move in the next 12 months

Exclusion Criteria:

1. Administration of rotavirus vaccine in the past
2. Presence of any illness requiring hospital referral (temporary exclusion)
3. Known case of immunodeficiency disease, known HIV positive
4. Known case of chronic gastroenteritis disease, chronic pulmonary disease, chronic renal disease, congenital heart disease
5. Any other conditions which in the judgment of the investigator warrant exclusion (e.g. no exclusion criteria but seems 'ill', investigators suspects neglect)
6. Diarrhea on the day of enrollment (temporary exclusion)
7. A known sensitivity or allergy to any components of the study vaccines.
8. Major congenital or genetic defect.
9. Has received any immunoglobulin therapy and/or blood products since birth.
10. History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study, at the discretion of the principal investigator.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5800 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of ROTAVAC5D | 14 days following the 3rd dose till the age of 1 year (12 months) + up to 14 days].
  Efficacy of ORV 116E in comparison to a placebo against moderate-severe rotavirus gastroenteritis defined as: episode of diarrhea (the passage of three or more loose or watery stools within a 24-hour period), with or without vomiting, that requires overnight hospitalization or rehydration therapy equivalent to World Health Organization (WHO) plan B (oral rehydration therapy) or plan C (intravenous rehydration therapy) in a medical facility such as a hospital, clinic, or supervised rural health care center

SECONDARY OUTCOMES:
Efficacy of Severe rotavirus gastroenteritis (>11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus occurring at least 14 days following the third dose | Till the age of 12 months + up to 14 days
  Severe rotavirus gastroenteritis (>11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus occurring at least 14 days following the third dose
To evaluate the efficacy of a ROTAVAC 5D against any severity of rotavirusgastroenteritis | Till the age of 1 year (12 months) + up to 14 days
  Any severity of gastroenteritis caused by non vaccine rotavirus from 14 days following the 3rd dose
To evaluate the efficacy of ROTAVAC 5D for rotavirus only gastroenteritis (absence of co-pathogens) | Throughout study period i.e.,30 months
  All primary and secondary endpoints indicated above for episodes that result positive only for rotavirus, and no other co-pathogen.
To evaluate the efficacy of a ROTAVAC 5D against any severity of gastroenteritis irrespective of etiology | till the age of 1 year (12 months) + up to 14 days
  Any severity of gastroenteritis irrespective of etiology from 14 days following the 3rd dose
To evaluate the efficacy of ROTAVAC 5D against severe (>11 on the 20 point Vesikari scoring scale) gastroenteritis irrespective of etiology | From 14 days following the 3rd dose till the age of 1 year (12months) + up to 14 days
  Severe (>11 on the 20 point Vesikari scoring scale) gastroenteritis irrespective of etiology f
To evaluate the intent to treat efficacy of ROTAVAC 5D against severe rotavirus gastroenteritis | till the age of 1 year (12 months) + up to 14 days
  Severe rotavirus gastroenteritis (≥11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus in the intent-to-treat population
Safety of the subjects during study period To assess the safety of ROTAVAC 5D for immediate and seven day adverse events, after all the 3 doses | From the day of vaccine administration to 7 days for all the three doses.
  During this period, will be solicited adverse events till 30 minutes after each vaccination (immediate solicited adverse events) and adverse events occurring within 7 days after each vaccination.
To assess the safety of ROTAVAC 5D for adverse events in the 4-week period following administration of each of the three doses of the vaccine/placebo | day 0 to 28 following each dose
  Unsolicited adverse events assessed from day 0 to 28 following each dose in comparison to a placebo will be assessed in a subset of subjects
To assess the safety of ROTAVAC 5D for SAEs,especially intussusception events occurring during the study period in all subjects | from day of 1st dose till the age of 1 year (12 months) + up to 14 days
  SAEs with a special focus on Intussusception events in comparison to a placebo will be assessed in all subjects throughout the study period.
Secondary Objectives (Immunogenicity) | Day 28 (+) 5 days after the third dose in comparison to baseline levels
  Immunogenicity rates after three doses of the ROTAVAC 5D in comparison to a placebo will be ascertained in approximately 150 subjects in each group assessed by fourfold rise in rotavirus-specific serum IgA antibody titers.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.V.Krishna Mohan, PhD, Study Director — Bharat Biotech International Limited
Locations (16):
- Chile (16):
  - Vacunatorio Mediped, Antofagasta
  - Vacunatorio Kinewen, Concepción
  - CESFAM Dr. Alejandro Gutierrez, Coyhaique
  - Hospital de Puerto Montt, Los Lagos
  - Hospital Base Osorno ,Av. Guillermo Buhler 1765, Osorno
  - CESFAM Puerto Aysen, Puerto Aisén
  - Centro de Salud Familiar CESFAM Rosita Renard, Santiago
  - Hospital de Carabineros, Santiago
  - Consultorio Dr. Alejandro del Rio, Santiago
  - Hospital de ninos Roberto del Rio, Santiago
  - CESFAM Esmeralda, Santiago
  - CESFAM Colina, Santiago
  - CESFAM Lo Barnechea, Santiago
  - Hospital Exequiel Gónzalez Cortés, Santiago
  - CESFAM Jean y Marie Thierry de Valparaíso, Valparaíso
  - Hospital Gustavo Fricke, Viña del Mar

IPD SHARING:
Plan to Share IPD: No